CLINICAL TRIAL: NCT06247683
Title: A Prospective, Non-comparative, Multicenter Trial to Confirm Safety and Performance of a New Multifocal IOL
Brief Title: Study to Confirm Safety and Performance of a New Multifocal IOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT ELANA 841P-BER-401-22
Record Dates: First submitted 2023-09-12; First posted 2024-02-08 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cataract Senile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- trifocal intraocular lens (Experimental): Bilateral Implantation of new trifocal intraocular lens
  Interventions: Device: trifocal intraocular lens

INTERVENTIONS:
Device: trifocal intraocular lens — cataract extraction and implantation of a posterior chamber trifocal intraocular lens

SUMMARY:
Prospective, non-comparative, multicenter study on medical device with 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient of any gender;
2. Patient with clinically significant bilateral age-related cataracts planned for phacoemulsification cataract extraction and eligible for implantation of a posterior chamber trifocal intraocular lens as determined by investigator's medical judgement;
3. Expected postoperative corrected distance visual acuity (CDVA) of 0.2 logMAR or better in both eyes as determined by investigator's medical judgement;
4. Preoperative corneal astigmatism <1.0 D;
5. Clear intraocular media other than cataract;
6. Requiring an IOL power within the available range of the investigational IOL (0.0 to +34.0 D, in 0.5 D increments);
7. Patient agrees to have surgery of the second eye performed between 1 day and 15 days after the surgery of the first eye.
8. Given written informed consent by patient;
9. Patient willing and able to comply with examination procedures and schedule for follow-up visits;

Exclusion Criteria:

1. Acute, chronic or uncontrolled systemic disease that could increase the operative risk or confound the outcome including but not limited to poorly controlled diabetes mellitus, active cancer treatment, mental illness, dementia, immunocompromised, connective tissue disease, clinically significant atopic disease, etc.;
2. Ocular condition that may predispose patient to future complications, per investigator's medical judgement, including but not limited to severe dry eye, anterior segment pathology, uncontrolled glaucoma, macular degeneration that would result in a visual acuity of 0.2 logMAR or worse during the study;
3. Clinically significant corneal abnormalities, including corneal dystrophy (epithelial, stromal or endothelial dystrophy), irregularity, inflammation or oedema as per Investigator's medical judgement; conditions including but not limited to keratitis, keratoconjunctivitis, kerato-uveitis, keratopathy, keratectasia;
4. Previous intraocular or corneal/refractive surgery that might confound the outcome of the investigation or increase the risk to the patient (including corneal transplants, removal of pterygium, and LASIK, LASEK, PRK, RK limbal relaxing incision etc.);
5. Use of and foreseeable use of systemic medications that may confound the outcome or increase the risk to the patient per investigator's medical judgement (e.g., steroids, Tamsulosin Hydrochloride or other medications including anticholinergics or alpha-adrenergic blocking agents with similar side effects [e.g. small pupil/floppy iris syndrome, lentodonesis], anti-metabolites, etc.);
6. Patients with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders, optic nerve atrophy etc.) or any other pathologies of the eye that are predicted to result in a visual acuity of 0.2 logMAR or worse during the study;
7. Patients with conditions that increase the risk of zonular rupture during cataract extraction procedure that may affect the stability of the IOL in the capsular bag (e.g. centration or tilt of the lens);
8. Planned concomitant ocular surgical procedure during cataract surgery or within the next 6 months (e.g. glaucoma surgery including implantation of MIGS, astigmatic correction surgery, penetrating keratoplasty, laser-assisted in situ keratomileusis);
9. Patients who are expected to require retinal laser treatment within the next 6 months per investigator's medical judgement;
10. Amblyopia, strabismus, single eye status;
11. Rubella, congenital, traumatic or complicated cataracts;
12. History of or current anterior or posterior segment inflammation, including but not limited to iritis or uveitis;
13. Microphthalmos or macrophthalmos;
14. Pupil abnormalities (e.g. aniridia, abnormal shaped pupils, non-reactive pupils);
15. Optic nerve atrophy;
16. Pseudoexfoliation;
17. Keratoconus or irregular astigmatism;
18. Inability to measure keratometry or biometry (including but not limited to cataract density, patient unable to focus for longer time etc.);
19. Pathologic miosis;
20. Pregnant, plan to become pregnant, lactating during the course of the investigation, or another condition with associated fluctuation of hormones that could lead to refractive changes;
21. Patients whose freedom is impaired by administrative or legal order;
22. Patients with nocturnal or glare prone occupational activities (e.g. taxi drivers)
23. Concurrent participation in another clinical investigation in the last 30 days.

    Intraoperative Exclusion criteria:
24. Need for additional iris manipulation (e.g., iris retractors);
25. Capsular fibrosis or opacities which might influence vision and the performance of the lens;
26. Inability to fixate the complete IOL stable in the capsular bag.

    * The eligibility criteria must be met in both eyes. If only one eye fulfils the criteria preoperatively, the patient cannot be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Monocular CDVA at 4 m in logMAR | 4-6 Month
  Comparison of mean CDVA to historical data of a monofocal control group

SECONDARY OUTCOMES:
Proportion of eyes with CDVA of 0.3 logMAR at 4 m | 4-6 Month

CONTACTS AND LOCATIONS:
Locations (11):
- Czechia (4):
  - Nemocnice Havlíčkův, Havlíčkův Brod
  - Fakultní nemocnice Královské Vinohrady, Prague
  - Oční Centrum Praha, Prague
  - Ústřední vojenská nemocnice - Vojenská fakultní nemocnice Praha, Prague
- Germany (3):
  - Augenklinik Ahaus GmbH & Co. KG, Ahaus
  - Augen-Medizinisches Versorgungszentrum, Landshut
  - AugenCentrum Rosenheim, Rosenheim
- Slovakia (4):
  - NeoVízia s.r.o., Bratislava
  - VESELY Očná Klinika, s.r.o., Bratislava
  - UVEA Klinika, s.r.o, Martin
  - Vidissimo s.r.o., Trenčín

REFERENCES:
- [Derived] Janekova A, Mojzis P, Nemcova I, Kacerik M, Vesely P, Hrckova L. Visual Outcomes of a New Hydrophobic Trifocal Intraocular Lens in Cataract Treatment: A Prospective Clinical Study. J Ophthalmol. 2025 Jul 24;2025:2662730. doi: 10.1155/joph/2662730. eCollection 2025. PMID 40746764